CLINICAL TRIAL: NCT07352956
Title: An 8-Week, Randomised, Controlled, Examiner-blind Clinical Study to Evaluate the Efficacy of a Stannous Fluoride Toothpaste for the Relief of Dentin Hypersensitivity in a Chinese Population
Brief Title: A Clinical Study to Evaluate the Effectiveness of an Test Toothpaste for the Relief of Dentin Hypersensitivity in a Chinese Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300265
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Toothpaste (Experimental): Participants will be instructed to brush the two test teeth first, then the whole mouth (all teeth) for at least 1-timed minute, twice daily (morning and evening) for 8 weeks. After brushing, participants will rinse once with 10 milliliter (ml) water using the measuring cup provided.
  Interventions: Drug: Test toothpaste
- Control Toothpaste (Other): Participants will be instructed to brush the whole mouth (all teeth) for 1-timed minute, twice daily (morning and evening) for 8 weeks. After brushing, rinse once with 10 ml water using the measuring cup provided.
  Interventions: Drug: Sodium fluoride toothpaste

INTERVENTIONS:
Drug: Test toothpaste — A toothpaste containing 0.454% SnF2.
  Arms: Test Toothpaste
Drug: Sodium fluoride toothpaste — A regular sodium fluoride toothpaste.
  Arms: Control Toothpaste

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of a 0.454 percent (%) weight/weight (w/w) stannous fluoride (SnF2) toothpaste in reducing dentin hypersensitivity (DH) to an evaporative (air) stimulus and tactile stimulus after 28 and 56 days twice daily brushing.

DETAILED DESCRIPTION:
This will be a single center, randomized, controlled, examiner-blind, 2-arm, stratified, parallel design clinical study in healthy male and female participants, aged 18-70, with self-reported and clinically confirmed DH in a Chinese population in a study design as per the Chinese Ministry of Health (MOH) Guidance. Sufficient participants will be screened so that approximately 100 participants (50 per group) will be stratified according to the maximum baseline Schiff sensitivity score of their two 'Test Teeth' and randomized to ensure approximately 90 evaluable participants (45 per group) complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent document confirming the participant has been informed of all pertinent aspects of the study and has given their written consent for study participation before any study procedures are performed.
* Participant is biologically male or female.
* Participant is 18 to 70 years of age at the time of signing the consent form.
* Participant is willing and able to comply with the study visit schedule, toothpaste usage instructions, lifestyle restrictions, and other study procedures.
* Participant is in good general, oral, and mental health, which in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in self-reported medical history, or upon oral examination that would impact their safety or wellbeing, or the outcomes of the study if they were to participate in the study, or affect their ability to understand and follow study requirements.
* Participant who is willing to receive reminders of appointments and videos reminding them on the brushing instructions.
* Participant must have a self-reported history of tooth sensitivity lasting more than 6 months but not more than 10 years and experience DH symptoms at least 'once a week' or more frequently.
* Participant must be in general oral health, with a minimum of 20 natural teeth.

Exclusion Criteria:

* Participant who is an employee of the study site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the study site otherwise supervised by the investigator; or a sponsor employee directly involved in the conduct of the study or a member of their immediate family.
* Participant who is participating in, or has participated in, other studies (including nonmedicinal studies) involving investigational product(s) within 8 weeks of Screening (Visit 1) or plans to participate in other studies (including non-medicinal studies) during this study.
* Participant who is participating in, or has participated in, a study evaluating a tooth desensitizing treatment within 8 weeks of Screening (Visit 1).
* Participant who is using or has used an oral care product indicated for DH relief within 8 weeks of Screening (Visit 1).
* Participant who has had a professional desensitizing treatment within 8 weeks of Screening (Visit 1).
* Participant with known or suspected intolerance or hypersensitivity to the study products or any of their stated ingredients (or closely related compounds).
* Participant who is unwilling or unable to comply with product usage instructions or Lifestyle Considerations as described in the protocol.
* Participant who habitually rinses with water during toothbrushing (self-reported at Screening (Visit 1), or those observed to rinse with water while brushing during the supervised brushing with the allocated toothpaste at screening (Visit 1) or baseline (Visit 2).
* Female participant who is pregnant or intending to become pregnant during the study (self-reported) or is breastfeeding.
* Participant with a recent history (within the last year) of alcohol and/or substance abuse.
* Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* Participant taking daily doses of medications or traditional herbal treatments which, in the opinion of the investigator or medically qualified designee, could interfere with their perception of pain.

  1. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, mood-altering and anti-inflammatory drugs.
  2. Examples of traditional herbal treatments include clove oil, olive oil or other treatments directly applied to the oral cavity for the treatment of oral health conditions.
* Participant taking daily doses of a medication which, in the opinion of the investigator or medically qualified designee, may cause xerostomia.
* Participant who needs antibiotic prophylaxis for dental procedures.
* Participant who has taken antibiotics within 2 weeks of screening (Visit 1) and Baseline visit (Visit 2) (during the acclimatization period).
* Participant who has had a professional or self-applied tooth bleaching procedure within 8 weeks of Screening (Visit 1).
* Participant who has had dental prophylaxis within 4 weeks of Screening (Visit 1).
* Participant who has had treatment for periodontal disease (including surgery) within 12 months of Screening (Visit 1).
* Participant who has had scaling or root planning within 3 months of Screening (Visit 1).
* Participant with a tongue or lip piercing.
* Participant with, in the opinion of the investigator or medically qualified designee, gross periodontal disease.
* Participant with evidence of gross intra-oral neglect or the need for extensive dental therapy.
* Participant with a fixed or removable partial prosthesis which, in the opinion of the investigator or medically qualified designee, would impact study outcomes.
* Participant with multiple dental implants which, in the opinion of the investigator or medically qualified designee, would impact study outcomes.
* Participant with fixed or removable orthodontic braces/bands or a fixed orthodontic retainer.
* Participant who is unable to provide appropriate responses to the VAS training exercise.
* Specific dentition exclusions for 'Test Teeth':

  1. Tooth with evidence of current or recent caries or reported treatment of decay within 12 months of Screening (Visit 1).
  2. Tooth with exposed dentin but with deep, defective or facial restorations.
  3. Tooth with full crown or veneer.
  4. Tooth adjacent to a bridge abutment or crown which, in the opinion of the investigator or medically qualified designee, would impact study outcomes.
  5. Sensitive tooth with contributing aetiologies other than EAR to exposed dentine.
  6. Sensitive tooth, in the opinion of the investigator or medically qualified designee, not expected to respond to treatment with an anti-sensitivity toothpaste.
* Participant who had previously been enrolled in this study.
* Any participant who, in the opinion of the investigator or medically qualified designee, was not expected to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Schiff Sensitivity Score at Day 56 | Baseline and Day 56
  Evaporative (air) sensitivity will be assessed by participant's response to an evaporative (air) stimulus after stimulation of 2 selected test teeth. Response of participant will be scored using Schiff sensitivity scale which ranges from 0-3, where 0=Does not respond to air stimulation; 1=Responds to air stimulus but does not request discontinuation of stimulus; 2=Responds to air stimulus and requests discontinuation or moves from stimulus; 3=Responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. Schiff sensitivity score= average score of the 2 'test teeth' identified at baseline. Change from baseline= Score at Day 56 minus baseline score. A decrease in Schiff sensitivity score indicates an improvement.
Change From Baseline in Tactile Threshold (grams [g]) at Day 56 | Baseline and Day 56
  The tactile sensitivity will be assessed by administrating a constant pressure using a Yeaple probe. The tactile threshold is the maximum pressure applied without the participant reporting pain or discomfort. The tactile threshold for 2 selected test teeth will be determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gives two consecutives 'yes' responses will be recorded as the tactile threshold. The greater the tactile threshold, the less sensitive the tooth. Tactile threshold= average value for the two 'test teeth' identified at baseline. Change from baseline= Score at Day 56 minus baseline score.

SECONDARY OUTCOMES:
Change From Baseline in Schiff Sensitivity Score at Day 56 (Test versus [vs] Control Toothpaste) | Baseline and Day 56
  Evaporative (air) sensitivity will be assessed by participant's response to an evaporative (air) stimulus after stimulation of 2 selected test teeth. Response of participant will be scored using Schiff sensitivity scale which ranges from 0-3, where 0=Does not respond to air stimulation; 1=Responds to air stimulus but does not request discontinuation of stimulus; 2=Responds to air stimulus and requests discontinuation or moves from stimulus; 3=Responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. Schiff sensitivity score= average score of the 2 'test teeth' identified at baseline. Change from baseline= Score at Day 56 minus baseline score. A decrease in Schiff sensitivity score indicates an improvement.
Change From Baseline in Tactile Threshold (g) at Day 56 (Test vs Control Toothpaste) | Baseline and Day 56
  The tactile sensitivity will be assessed by administrating a constant pressure using a Yeaple probe. The tactile threshold is the maximum pressure applied without the participant reporting pain or discomfort. The tactile threshold for 2 selected test teeth will be determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gives two consecutives 'yes' responses will be recorded as the tactile threshold. The greater the tactile threshold, the less sensitive the tooth. Tactile threshold= average value for the two 'test teeth' identified at baseline. Change from baseline= Score at Day 56 minus baseline score.
Change From Baseline in Schiff Sensitivity Score at Day 28 | Baseline and Day 28
  Evaporative (air) sensitivity will be assessed by participant's response to an evaporative (air) stimulus after stimulation of 2 selected test teeth. Response of participant will be scored using Schiff sensitivity scale which ranges from 0-3, where 0=Does not respond to air stimulation; 1=Responds to air stimulus but does not request discontinuation of stimulus; 2=Responds to air stimulus and requests discontinuation or moves from stimulus; 3=Responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. Schiff sensitivity score= average score of the 2 'test teeth' identified at baseline. Change from baseline= Score at Day 28 minus baseline score. A decrease in Schiff sensitivity score indicates an improvement.
Change From Baseline in Tactile Threshold (g) at Day 28 | Baseline and Day 28
  The tactile sensitivity will be assessed by administrating a constant pressure using a Yeaple probe. The tactile threshold is the maximum pressure applied without the participant reporting pain or discomfort. The tactile threshold for 2 selected test teeth will be determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gives two consecutives 'yes' responses will be recorded as the tactile threshold. The greater the tactile threshold, the less sensitive the tooth. Tactile threshold= average value for the two 'test teeth' identified at baseline. Change from baseline= Score at Day 28 minus baseline score.
Change From Baseline in (Visual Analogue Scale) VAS Scores at Day 28 and 56 | Baseline, Day 28 and Day 56
  Evaporative (air) sensitivity will be assessed by participant's response to an evaporative (air) stimulus after stimulation of 2 selected test teeth. Response of participant will be scored using Schiff sensitivity scale which ranges from 0-3, where 0=Does not respond to air stimulation; 1=Responds to air stimulus but does not request discontinuation of stimulus; 2=Responds to air stimulus and requests discontinuation or moves from stimulus; 3=Responds to stimulus, considers stimulus to be painful and requests discontinuation of the stimulus. Participants then rated the intensity of their response to the evaporative (air) stimulus using a 100 millimeter (mm) VAS with scores ranging from 0 mm (No discomfort) to 100 mm (extreme discomfort; worst imaginable). Higher score indicated worse outcome (higher sensitivity). Change from baseline will be calculated by subtracting Baseline value from the value at the indicated timepoints.

CONTACTS AND LOCATIONS:
Locations (1):
- West China School/Hospital of Stomatology, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.